CLINICAL TRIAL: NCT01724762
Title: Evaluation of the Efficacy of Nursing Orientation to Reduce the Anxiety of Patients With Acute Coronary Syndrome Undergoing Bed Bath
Brief Title: Efficacy of Nursing Orientation to Reduce the Anxiety of Patients Undergoing Bed Bath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Juliana de Lima Lopes, Master Degree, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UNIFESP0447
Record Dates: First submitted 2012-11-06; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Baths; Anxiety; Acute Coronary Syndrome; Education, Nursing
MeSH Terms: conditions — Acute Coronary Syndrome; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nursing orientation (Experimental): Patients who received nursing orientation and read the informative manual concerning bed bath
  Interventions: Other: Nursing Orientation

INTERVENTIONS:
Other: Nursing Orientation — * Control group: patients who did not read the informative manual concerning bed bath and received only the unit's routine information
  * Intervention group: patients who received nursing orientation and read the informative manual concerning bed bath

SUMMARY:
This study's general objective was to evaluate the efficacy of nursing orientation to reduce the anxiety of patients with acute coronary syndrome undergoing bed bath. The specific objectives included: the development and validation of an informative manual concerning bed bath; correlation of physiological variables (systolic and diastolic blood pressure and heart and respiratory rate) with the patients' state anxiety; correlation of antecedent variables (age, gender, cardiovascular risk factor, use of beta blockers, trait anxiety, depression, prior hospitalization, prior experience with bed baths, the patients' preference for a female or male professional to perform the bath, pain, fear, and embarrassment) with the patients' state anxiety.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome present many physiological and psychological changes, especially anxiety, which can be more intense when the patient expects or experiences certain procedures, such as bed bath. The association of anxiety and acute myocardial infarction has shown negative impact on the prognosis of these patients. The anxiety causes activation of the sympathetic nervous system by increasing cardiac contractility, blood pressure, heart rate and oxygen consumption, worsening disease progression. Thus, minimizing the effects of patients' anxiety in the face of various nursing procedures is essential to quality care. The anxiety can be reduced using medications and/or nursing orientation.

This study was conducted in the Coronary Care Units, Brazilian Heart Institute. The study was divided into two phases. The first comprised the development and validation of an informative manual by nurses and patients. The manual was developed by the researchers and then submitted to validation by five nursing professors from the field of nursing fundamentals and five nurses with experience in coronary care units. The Delphi Technique was used to validate the manual in this phase. After validation by nurses, the manual was validated by 35 patients hospitalized in the coronary care unit who experienced bed bath at least once. A score above 4 should be achieved for the manual to be considered comprehensible and validated by patients. The statistical analysis at this phase was performed through the Wilcoxon rank-sum test and percentage of score 5 with its confidence interval. The study's second phase comprised assessment of the efficacy of nursing orientation to reduce the anxiety of patients with acute coronary syndrome undergoing bed baths. The sample population was composed of 120 patients with acute coronary syndrome hospitalized in coronary care units divided into two groups: control group (patients who did not read the informative manual concerning bed bath and received only the unit's routine information) and the intervention group (patients who received nursing orientation and read the informative manual concerning bed bath). The STAI-state was used to assess anxiety. It was applied immediately after informing the patients about the bed bath, immediately after orientation (intervention group) or immediately after the unit's routine information (control group), and immediately after the bath.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute coronary syndrome Killip 1
* Patients who were undergoing the bed bath for the first time in the current hospitalization
* Literate and at least 4 years of study
* Patients with age less than 75 years
* Patients who agreed to participate

Exclusion Criteria:

* Patients with vascular diseases or arteriovenous fistulas in the left arm
* Situations that could influence patients' anxiety and / or vital signs (arrhythmias such as ventricular tachycardia, second or third-degree atrioventricular block ; ischemic pain before, during or after bath; patients with Killip 2, 3 and 4; invasive procedures on the day of data collection, such as catheterization and surgery, and use of benzodiazepines and / or anxiolytics
* Situations in which patients were not able to complete the questionnaires (altered level of consciousness, visual impairment and / or patients who could not read and / or write)
* Situations in which the patient requested information about bed bath, previously the beginning of the evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
STAI-state | Participants were followed for the duration of hospital stay, an average of 2 weeks
  The STAI-state was applied immediately after informing the patients about the bed bath, immediately after orientation (intervention group) or immediately after the unit's routine information (control group), and immediately after the bath.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana L Lopes, Ms, Principal Investigator — Federal University of São Paulo; Alba LB Barros, PhD, Study Director — Federal University of São Paulo; Luiz A Nogueira-Martins, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Lopes Jde L, Nogueira-Martins LA, Goncalves MA, de Barros AL. Comparing levels of anxiety during bed and shower baths in patients with acute myocardial infarction. Rev Lat Am Enfermagem. 2010 Mar-Apr;18(2):217-23. doi: 10.1590/s0104-11692010000200012. PMID 20549121
- [Result] Barsevick A, Llewellyn J. A comparison of the anxiety-reducing potential of two techniques of bathing. Nurs Res. 1982 Jan-Feb;31(1):22-7. PMID 6922456
- [Result] Tel H, Tel H. The effect of individualized education on the transfer anxiety of patients with myocardial infarction and their families. Heart Lung. 2006 Mar-Apr;35(2):101-7. doi: 10.1016/j.hrtlng.2005.09.001. PMID 16543038
- See also: American Heart Association — http://www.heart.org/HEARTORG/